CLINICAL TRIAL: NCT06647394
Title: Efficacy of Application of Myriad Matrix to Split Thickness Skin Graft Sites
Status: Withdrawn | Type: Observational
Why Stopped: The study never opened or enrolled any subjects.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Benjamin Greene, Associate Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300013305; UAB (Other: UAB)
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Skin Grafts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Matrix Dressing — extracellular matrix dressing soaked in 4% topical lidocaine to the skin graft donor site

SUMMARY:
To determine if application of Myriad Matrix to split thickness skin graft donor sites improves post-operative pain and appearance of the wound.

DETAILED DESCRIPTION:
In the head and neck practice at UAB, split thickness skin grafts are a commonly used procedure for simple reconstruction. The standard dressing for donor sites is a strip of vaseline gauze which remains on the site the wound dries, and the gauze eventually falls off. Post operative pain and poor wound healing is a well established complication of the donor site, and various methods have been studied in an attempt to reduce these complications for patients in the post operative period. (1, 2, 3)

Myriad matrix is an engineered extracellular matrix (Ovine Forestomach Matrix) used for soft issue repair in complex wounds. This has been sporadically used by some of the faculty members at UAB for split thickness skin graft donor site dressings with anectodal improvement in pain and healing, though this has not yet been studied to our knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and over who are undergoing a split thickness skin graft at UAB.

Exclusion Criteria:

* Patients who are not planned to undergo a split thickness skin graft or who are unable or do not plan to attend follow up appointments will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing a split thickness skin graft
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Pain Improvement | 48 hours, 2 weeks, 4-6 weeks post operative visit
  patients will rate pain level at donor site
Wound Healing | 2 weeks and 4-6 weeks post operative visit
  Patients will rate appearance of would using the scar-Q questionnaire

IPD SHARING:
Plan to Share IPD: No